CLINICAL TRIAL: NCT04235062
Title: NATriuretic Response to Expansion and dIUretics in huMans With Heart Failure
Acronym: NATRIUM-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Momentum Research, Inc. (Industry)
Collaborators: Saint-Louis-Lariboisière University Hospitals (Unknown); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHF201901
Record Dates: First submitted 2020-01-15; First posted 2020-01-21 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Sodium Chloride; Calcium Chloride; Potassium Chloride; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluid Expansion and Diuretic Challenge (Experimental): Subject receive intravenous infusion of Ringer's (8.6 g/L sodium chloride, 0.33 g/L calcium chloride, 0.3 g/L potassium chloride) solution, followed by diuretic challenge with 40mg Furosemide intravenous bolus.
  Interventions: Drug: Ringer's (8.6 g/L sodium chloride, 0.33 g/L calcium chloride, 0.3 g/L potassium chloride) Solution; Drug: Intravenous Bolus Furosemide

INTERVENTIONS:
Drug: Ringer's (8.6 g/L sodium chloride, 0.33 g/L calcium chloride, 0.3 g/L potassium chloride) Solution — A 2-hour of infusion of Ringer's (8.6 g/L sodium chloride, 0.33 g/L calcium chloride, 0.3 g/L potassium chloride) solution will be given following completion of the first 3-hour urine collection period: 0.5 liter infused over 10 min followed by 0.5 liter infused over 1 hour 50 minutes.
  Other Names: Intravascular fluid expansion
Drug: Intravenous Bolus Furosemide — Following completion of the second 3-hour urine collection period and after the second set of blood and urine samples are obtained, 40 mg of furosemide will be given as an IV bolus.
  Other Names: Loop diuretic administration

SUMMARY:
NATRIUM-HF is a multicenter, non-randomized, pre-post intervention study designed to assess renal response to intravascular fluid expansion and diuretics after sacubitril/valsartan (Entresto®) in euvolemic heart failure patients with reduced ejection fraction. Approximately 230 eligible patients will attend one visit prior to and visits 2 and 3 months after starting Entresto®. At each visit, the patient's responses to extravascular fluid expansion with Ringer's solution and to a loop diuretic bolus will be measured. Biomarkers measured in blood and urine samples will include natriuretic peptides (NP) B-type NP (BNP) and N-terminal proBNP (NT-proBNP), NP fragments, neprilysin activity and concentration, and other biomarkers related to heart failure.

DETAILED DESCRIPTION:
NATRIUM-HF is a multicenter, non-randomized, pre-post intervention study designed to assess renal response to intravascular fluid expansion and diuretics after sacubitril/valsartan (Entresto®) in euvolemic heart failure patients with reduced ejection fraction.

Ambulatory patients with HFrEF who remain symptomatic despite optimal treatment for more than 3 months with an ACEi or ARB, a beta-blocker and a mineralocorticoid receptor antagonist (MRA) for whom sacubitril/valsartan is indicated and is about to be initiated will be enrolled. Approximately 230 patients will attend three outpatient visits: before, and 2 months and 3 months after initiation of, or switch from treatment with angiotensin-converting-enzyme inhibitor (ACEi) or angiotensin II receptor blocker (ARB) to, oral treatment with the angiotensin receptor-neprilysin inhibitor (ARNi) sacubitril/valsartan (Entresto®). Patient's responses to fluid expansion and diuretic administration will be assessed at each study visit.

The same procedures will be followed at each visit. First, baseline vital signs, clinical assessments (dyspnea score, jugular vein distension, peripheral edema score, pulmonary rales), and blood samples will be obtained. Urine will be collected over a period of 3 hours and urine samples will be obtained from the collected urine at the end of the 3-hour collection period, and vital signs and clinical assessments will be obtained.

This will be followed by an infusion of 0.5 liter Ringer's (8.6 g/L sodium chloride, 0.33 g/L calcium chloride, 0.3 g/L potassium chloride) solution infused in 10 min followed by an infusion of 0.5 liter over 1 hour 50 minutes. Of note 1liter Ringer's contains 8.6 g or 374 mmol of sodium. 1 hour after the end of the infusion, clinical assessments (dyspnea score, jugular vein distension, peripheral edema score, pulmonary rales) and blood samples will be obtained. Urine will be collected over a period of 3 hours and urine samples will be obtained from the collected urine at the end of the 3-hour collection period.

After the second set of blood and urine samples are obtained, 40 mg of furosemide will be given IV and blood samples will be obtained thereafter hourly for 3 hours. Urine will be collected over a period of 3 hours and urine samples will be obtained from the collected urine at the end of the 3-hour collection period, and vital signs and clinical assessments will be obtained.

Biomarkers measured in blood and urine samples will include natriuretic peptides (NP) B-type NP (BNP) and N-terminal proBNP (NT-proBNP), NP fragments, neprilysin activity and concentration, and other biomarkers related to heart failure.

The aim of NATRIUM-HF is to assess the change in natriuretic response to intravascular fluid expansion and diuretics in euvolemic patients with heart failure and reduced ejection fraction (HFrEF) after initiation of, or switch from ACEi/ARB to, sacubitril/valsartan (Entresto®) therapy.

ELIGIBILITY:
Inclusion criteria:

1. Male or female patients ≥ 18 and < 80 years of age.
2. Ambulatory patients with a diagnosis of stable NYHA class II heart failure with left ventricular ejection fraction <40 %, for whom sacubitril/valsartan (Entresto®) is indicated as recommended by ESC guidelines and are about to be switched to Entresto® therapy.
3. Stable oral doses of ACEi or ARB, beta-blocker, mineralocorticoid antagonist (MRA), and loop diuretic (up to 120 mg daily furosemide or equivalent*) for > 3 months prior to Screening, except where intolerance or contraindication documented.
4. Stable HF without any recent exacerbation of symptoms and/or signs of HF, admission for HF, unplanned clinic visit or emergency service visit for HF or need for significant up titration or new administration of oral or IV diuretics, renin-angiotensin system (RAAS) blockers (including ACEi, ARB, and/or MRA) and/or beta blockers for > 3 months.
5. Euvolemia as defined by no signs of congestion (pulmonary rales or >1+ peripheral edema) by physical examination.
6. Written informed consent to participate in the study.
7. Ability to comply with all study requirements, without major morbidities compromising the patient's ability to participate and understand the study for 90 days.

Exclusion criteria:

1. Significant pulmonary disease contributing substantially to the patients' dyspnea such as FEV1< 1 liter or need for chronic steroid therapy.
2. Myocardial infarction, unstable angina, ICD or CRT implantation, or cardiac surgery, including percutaneous transluminal coronary intervention, within past 3 months.
3. History of heart transplant or on a transplant list, or using or planned to be implanted with a ventricular assist device.
4. Sustained ventricular arrhythmia with syncopal episodes within past 3 months that is untreated.
5. Presence of any hemodynamically significant valvular stenosis or regurgitation, except mitral or tricuspid regurgitation secondary to left ventricular dilatation. Presence of hemodynamically significant obstructive lesions of left ventricular outflow tract.
6. Stroke or TIA within the past 3 months
7. Primary liver disease considered to be life threatening.
8. Any episode of symptomatic hypotension within 3 months prior to screening.
9. Known history of angioedema with ACEi or ARB use, or history of hereditary or idiopathic angioedema.
10. Coagulation or bleeding disorder.
11. Systolic blood pressure < 100 mmHg.
12. Serum sodium > 146 mEq/L (146 mmol/L).
13. Serum potassium > 5.2 mEq/L (5.2 mmol/L) or < 3.5 mEq/L (3.5 mmol/L).
14. Renal disease or eGFR < 30 ml/min/1.73m2 (as measured by the simplified MDRD formula).
15. Ultrafiltration or dialysis within 3 months prior to Screening.
16. Hypersensitivity to sacubitril, valsartan, or any of the excipients in Entresto®; or hypersensitivity to furosemide.
17. History or presence of any other diseases (i.e. including malignancies) with a life expectancy of < 3 months.
18. Participation in any CHF trial or any investigational drug or device study within the 30 days prior to Screening.
19. History of noncompliance to medical regimens and patients who are considered potentially unreliable.
20. Pregnant or nursing (lactating) women.
21. Active infection based on abnormal temperature and elevated WBC count.
22. Receipt of blood transfusion within 3 months prior to Screening.
23. Current use of any drug containing a direct renin inhibitor (aliskiren) or neprilysin inhibitor (sacubitril).

    * Equivalent oral loop diuretic doses will be considered as 1 mg bumetanide=20 mg torsemide=80 mg furosemide

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Natriuretic response to intravascular volume expansion | 2 and 3 months
  The average change in natriuretic response to intravascular volume expansion from before to 2 and 3 months after initiation of sacubitril/valsartan therapy. Natriuretic response is defined as the cumulative sodium excretion over the 3 hours of intravascular volume expansion and follow up.
Natriuretic response to IV diuretic administration | 2 and 3 months
  The average change in cumulative natriuresis during the first 3 h following the bolus IV furosemide administration from before to 2 and 3 months after initiation of sacubitril/valsartan therapy.

SECONDARY OUTCOMES:
Natriuretic peptide (NP) response to intravascular volume expansion | 2 and 3 months
  Change from from before to 2 and 3 months after initiation of sacubitril/valsartan therapy in the average change over the 2-hour Ringer's infusion and follow up in plasma NP levels from just prior to the start of the infusion.
Natriuretic peptide response to IV diuretic administration | 2 and 3 months
  Change from before to 2 and 3 months after initiation of sacubitril/valsartan therapy in the average change in NP level from the end of the Ringer's infusion to 3 hours following the bolus IV furosemide administration
Diuretic response | 2 and 3 months
  Change from before to 2 and 3 months after initiation of sacubitril/valsartan therapy in the urine volume excreted over the 3 hours following the bolus IV furosemide administration
4. Changes in dyspnea as measured by a 1-10 scale in response to intravascular fluid expansion, and diuretic administration | 2 and 3 months
  Change from before to 2 and 3 months after initiation of sacubitril/valsartan therapy in the average change from just prior to the Ringer's infusion start to one hour following the 2-hour Ringer's infusion and from just prior to the IV bolus furosemide administration to 3 hours following the bolus IV furosemide administration

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Mebazaa, MD PhD FESC, Principal Investigator — Hôpitaux Universitaires Saint-Louis-Lariboisière
Locations (13):
- Armenia (4):
  - Erebouni Medical Center CJSC, Yerevan
  - Institute of Cardiology named after L.A. Hovhannisyan, Yerevan
  - Nairi Medical Center, Yerevan
  - Yerevan State Medical University, Yerevan
- Bosnia and Herzegovina (2):
  - University Clinical Center Republic of Srpska, Banja Luka Department of Cardiology, Banja Luka
  - University Clinical Center Mostar, Mostar
- Russia (7):
  - Regional budget Healthcare Institution "Cardiological dispensary", Ivanovo
  - Moscow State Budgetary Institution of Healthcare of Moscow "City Clinical Hospital named after V.V. Vinogradov of the Department of Healthcare of Moscow", Moscow
  - State Budgetary Healthcare Institution of Moscow "City clinical hospital #51 of the Department of Healthcare of Moscow", Moscow
  - State Budgetary Healthcare Institution of Moscow "City Clinical Hospital named after V.V. Veresaev of the Department of Healthcare of Moscow", Moscow
  - State Budgetary Healthcare Institution of Moscow "Moscow City Clinical Hospital named after V.M. Buyanov" of the Department of Healthcare of Moscow", Moscow
  - MedFort LLC, Saint Petersburg
  - State Budgetary Healthcare Institution of Vladimir region "Vladimir City Hospital # 4", Vladimir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McMurray JJ, Packer M, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile MR; PARADIGM-HF Investigators and Committees. Angiotensin-neprilysin inhibition versus enalapril in heart failure. N Engl J Med. 2014 Sep 11;371(11):993-1004. doi: 10.1056/NEJMoa1409077. Epub 2014 Aug 30. PMID 25176015
- [Background] Nijst P, Verbrugge FH, Martens P, Dupont M, Tang WHW, Mullens W. Renal response to intravascular volume expansion in euvolemic heart failure patients with reduced ejection fraction: Mechanistic insights and clinical implications. Int J Cardiol. 2017 Sep 15;243:318-325. doi: 10.1016/j.ijcard.2017.05.041. Epub 2017 May 14. PMID 28545850
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JG, Coats AJ, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GM, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; Authors/Task Force Members; Document Reviewers. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2016 Aug;18(8):891-975. doi: 10.1002/ejhf.592. Epub 2016 May 20. No abstract available. PMID 27207191
- [Background] Tuttolomondo A, Pinto A, Di Raimondo D, Corrao S, Di Sciacca R, Scaglione R, Caruso C, Licata G. Changes in natriuretic peptide and cytokine plasma levels in patients with heart failure, after treatment with high dose of furosemide plus hypertonic saline solution (HSS) and after a saline loading. Nutr Metab Cardiovasc Dis. 2011 May;21(5):372-9. doi: 10.1016/j.numecd.2009.10.014. Epub 2010 Mar 25. PMID 20346637